CLINICAL TRIAL: NCT07234760
Title: ex Vivo Study of Liposomes Loaded With Everolimus in Chronic Lung Allograft Disfunction
Acronym: ELIT
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Mirko Belliato, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: ELIT
Record Dates: First submitted 2025-09-22; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-09

CONDITIONS: Bronchiolitis Obliterans Syndrome (BOS)
Keywords: liposome
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — PCLS (precision cut lung slices); Lung fibroblast
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BOS
  Interventions: Device: Liposomes

INTERVENTIONS:
Device: Liposomes — 1. LIP(ev)-HA400kDa on lung fibroblasts derived from Broncoalvealar lavage of BOS affected patients checking key elements involved in pro-fibrotic signals in order to understand if our nanovehicle could modulate process basing fibrotic lesions production.
  2. LIP(ev)-HA400kDa and fluorescent LIP-HA400kDa in PCLSs from explanted lungs by BOS patients in order to assess the cellular distribution of LIP-HA400kDa and the effect

SUMMARY:
Patients subjected to lung transplantation develop acute rejection or chronic rejection with an incidence of 45% after the first year. The major clinical phenotype of chronic rejection is bronchiolitis obliterans syndrome (BOS), which cause an establishment of chronic lung inflammation status with an aberrant proliferation of myofibroblasts leading to fibrotic obstruction of small airways. The therapeutic regimen available for BOS patients is still scarce and is not able to revert the disease. This project aims to design a new targeted therapy based on nanoparticles that can deliver drug directly inside lungs by aerosol administration to revert BOS.

By this project will be exploit a liposomes preparation synthesized modifying surface with hyaluronic acid (HA), the physiologic ligand of CD44, a glycoprotein overexpressed by myofibroblasts forming fibrotic lesions. These targeted liposomes are loaded with everolimus (LIP(ev)-HA400kDa), a mTOR inhibitors already used for BOS patients but with significant side effects leading to a discontinuation of therapy. Loading everolimus inside liposomes allows the administration of drug directly to the lungs and decreases its side effects.

LIP(ev)-HA400kDa will be tested on different experimental settings: in vitro, ex vivo, in vivo. This approach will allow us to have a complete observation regarding the effects and the distribution of liposomes preparation, from the modulation of their specific targeting (myofibroblasts) by in vitro experiments, the analysis of LIP(ev)-HA400kDa behavior on human lung tissues and, finally, their ability to revert BOS in animal model.

Results obtained with this project will open to a new therapeutic option for BOS affected patients, the first therapy that can revert the disease prolonging the long-term survival of patients.

DETAILED DESCRIPTION:
LFs will be isolated from BAL of BOS-affected or subjected to TX. After isolation and culture, LFs will be incubated with LIP(ev)-HA400kDa, LIP(ev) and everolimus alone, comparing the effect to control cells. At the end of the incubation, we will collect supernatants and proteins of lysed cells. Proteins extracted will be quantified and western blot will be performed to assess the expression of collagen I, fibronectin and laminin. Regarding supernatants we will evaluate cytokines concentration, in particular: IL6, IL8, TGF-beta and IL10.

LIP-HA400kDa fluorescently labelled will be incubated onto PCLSs derived from BOS explanted lungs comparing their distribution with LIP-PEG, using confocal microscopy. Moreover, using LIP(ev)-HA400kDa, LIP(ev) and everolimus alone we will assess general toxicity on PCLSs using LDH assay and cell proliferation with Ki67 expression at different time points. We will also assess the release of cytokines involved in pro-inflammation and pro-fibrotic processes.

ELIGIBILITY:
Inclusion Criteria:

- BOS/subjected to TX patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: BOS affected patients
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2022-03-19 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
TGF-beta's levels in BAL cells | from 24 hours to 72 hours of treatment
  Comparison of TGF-beta levels in BAL cells in cells alone, nanoparticles alone, nanoparticles with drug delivery, and drug alone

SECONDARY OUTCOMES:
cytokine's levels in BAL's cells | from 24 hours to 72 hours of treatment
  Compare IL6, IL8, and IL10 levels in BAL cells in the four conditions.
cytokines and TGF-beta's levels released by PCLSs | from 24 hours to 72 hours of treatment
  Compare the levels of cytokines IL6, IL8, IL10, and TGF-beta released by PCLSs derived from explanted lungs and evaluate toxicity and cell proliferation.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kelsh SE, Girgis R, Dickinson M, McDermott JK. Everolimus Use for Intolerance or Failure of Baseline Immunosuppression in Adult Heart and Lung Transplantation. Ann Transplant. 2018 Oct 23;23:744-750. doi: 10.12659/AOT.910952. PMID 30348935
- [Background] Lopez P, Kohler S, Dimri S. Interstitial Lung Disease Associated with mTOR Inhibitors in Solid Organ Transplant Recipients: Results from a Large Phase III Clinical Trial Program of Everolimus and Review of the Literature. J Transplant. 2014;2014:305931. doi: 10.1155/2014/305931. Epub 2014 Dec 18. PMID 25580277
- [Background] Klawitter J, Nashan B, Christians U. Everolimus and sirolimus in transplantation-related but different. Expert Opin Drug Saf. 2015 Jul;14(7):1055-70. doi: 10.1517/14740338.2015.1040388. Epub 2015 Apr 26. PMID 25912929
- [Background] Chung PA, Dilling DF. Immunosuppressive strategies in lung transplantation. Ann Transl Med. 2020 Mar;8(6):409. doi: 10.21037/atm.2019.12.117. PMID 32355853
- [Background] Tissot A, Danger R, Claustre J, Magnan A, Brouard S. Early Identification of Chronic Lung Allograft Dysfunction: The Need of Biomarkers. Front Immunol. 2019 Jul 17;10:1681. doi: 10.3389/fimmu.2019.01681. eCollection 2019. PMID 31379869
- [Background] Verleden GM, Glanville AR, Lease ED, Fisher AJ, Calabrese F, Corris PA, Ensor CR, Gottlieb J, Hachem RR, Lama V, Martinu T, Neil DAH, Singer LG, Snell G, Vos R. Chronic lung allograft dysfunction: Definition, diagnostic criteria, and approaches to treatment-A consensus report from the Pulmonary Council of the ISHLT. J Heart Lung Transplant. 2019 May;38(5):493-503. doi: 10.1016/j.healun.2019.03.009. Epub 2019 Apr 3. No abstract available. PMID 30962148
- [Background] Mrad A, Chakraborty RK. Lung Transplant Rejection. 2022 Sep 26. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK564391/ PMID 33232061